CLINICAL TRIAL: NCT00432952
Title: Acute Single Meal Effects of Trout on Cardiovascular Risk Markers and Plasma Proteome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Institute of Fisheries Research (Other)
Responsible Party: Associate profesor Lotte lauritzen, Dept. of Human Nutrtion
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: M186
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome
Keywords: Cardiovascular Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

INTERVENTIONS:
Behavioral: Intake of rainbow trout from different feeding conditions versus a control poultry meal

SUMMARY:
The acute effects of farmed rainbow trout, fed by various feeds versus a control meal with poultry meat on cardiovascular risk markers and plasma protein expression are investigated.

The hypotheses of the study are that if the feed are changed from a marine origin to primarily a vegetable origin the content of long chain n-3 poly unsaturated fatty acids (n-3 PUFA) will decrease in the meat and thus possibly result in a decreased effect on health. Furthermore, the feed of the trouts are also expected to give rise to differences in the human plasma protein profile and fatty acid composition after consumption, which could be associated with physiological effects.

DETAILED DESCRIPTION:
In a controlled, single blinded human single meal study the acute effects of farmed rainbow trout, fed by various feeds versus a control meal with poultry meat on cardiovascular risk markers and plasma protein expression are investigated. 6 healthy men, age 40-70, will be randomized to trout fed on only vegetable, only marine and a mix of different compositions of vegetable and marine feeds. Outcome variables are blood pressure, pulse wave analyse, pulse wave velocity, plasma protein profile, and plasma triglycerides.

The hypotheses of the study are that if the feed are changed from a marine origin to primarily a vegetable origin the content of long chain n-3 poly unsaturated fatty acids (n-3 PUFA) will decrease in the meat and thus possibly result in a decreased effect on health. Furthermore, the feed of the trouts are also expected to give rise to differences in the human plasma protein profile and fatty acid composition after consumption, which could be associated with physiological effects.

ELIGIBILITY:
Inclusion Criteria:

* Non regular smokers
* Body Mass Index (18.5-30 kg/m2)
* Able to eat fish

Exclusion Criteria:

* Exercise >10 h/week
* Chronical diseases (eg. cardiovascular and diabetes)
* Regular medication
* Fish oil supplementation
* Blood donation 2 month prior or during participation
* Above maximum recommended alcohol intake
* Blood pressure >160/100 mm Hg

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
plasma protein expression
Blood Pressure
Pulse Wave Analysis
Pulse wave Velocity

SECONDARY OUTCOMES:
Plasma Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, Ph.D, Principal Investigator — University of Copenhagen
Locations (1):
- Institute of Human Nutrition, University of Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Rentsch ML, Lametsch R, Bugel S, Jessen F, Lauritzen L. The effects of eating marine- or vegetable-fed farmed trout on the human plasma proteome profiles of healthy men. Br J Nutr. 2015 Feb 28;113(4):699-707. doi: 10.1017/S0007114514004152. Epub 2015 Jan 27. PMID 25622825